CLINICAL TRIAL: NCT01000779
Title: Comparison of Endoscopic Variceal Ligation (EVL) and Propranolol in Secondary Prophylaxis of Variceal Bleeding in Patients With Non Cirrhotic Portal Hypertension (NCPH): A Prospective Randomized Controlled Trial
Brief Title: Comparison of Endoscopic Variceal Ligation (EVL) With Propranolol in Non Cirrhotic Portal Hypertension (NCPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Shiv K Sarin, G.B. Pant Hospital, New Delhi, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NG001
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2009-10

CONDITIONS: Non Cirrhotic Portal Hypertension
Keywords: Non Cirrhotic Portal Hypertension, secondary prophylaxis
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic Variceal Ligation (Active Comparator): endoscopic therapy to obliterate varices
  Interventions: Device: multi band ligator for esophageal varices
- Propranolol (Active Comparator): drugs to decrease portal pressure
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — upto 320mg/day maximum
  Arms: Propranolol
Device: multi band ligator for esophageal varices — to obliterate esophageal varices
  Arms: Endoscopic Variceal Ligation

SUMMARY:
Background: Variceal bleeding is a major cause of morbidity and mortality in patients with Non Cirrhotic Portal Hypertension (NCPH). Beta blockers (BB) and endoscopic variceal ligation (EVL) have been used to prevent rebleeding in these patients, largely based on data from cirrhotic patients. Endotherapy in the form of EST has been well studied in preventing rebleed in patients with NCPH. Initial studies showed that EST significantly reduced the rebleeding rate in patients of NCPH. Data from these studies suggests a rebleed rate of approximately 25% at 2yr and 35% at 5 years.

Beta blockers have been found to be quite effective in both primary as well as secondary prophylaxis of variceal bleeding in cirrhotic and are accepted mode of treatment. In contrast to liver cirrhosis, published data on the effect of beta blocker therapy on NCPH are scanty. Animal data and human data suggests that beta blockers reduce portal pressure in patients with NCPH. In two placebo controlled trials of propranolol on secondary prophylaxis of variceal bleeding in non cirrhotic patients. both studies demonstrated the efficacy of propranolol in decreasing rebleed rate. However, no comparisons hae been made with EVL till date.

Hypothesis: The investigators hypothesis that In patients with NCPH, treatment with beta blockers will lead to reduction in portal pressure and decrease in portosystemic shunting leading to reduction in variceal rebleeding Aim of the study: Aim: To compare the efficacy and safety of Propranolol and EVL in the prevention of variceal rebleeding in patients with NCPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Non Cirrhotic Portal Hypertension (NCPH) presenting to our Liver Diseases Follow-up Clinic with history of hemetemesis and/or malena within the past 6 weeks and proven to have esophageal varices as the bleeding source on upper GI endoscopy

Exclusion Criteria:

* A history of surgery for portal hypertension
* Patients already on a EST, EVL, or glue injection program before presenting to our hospital
* Patients already on beta blockers for primary prophylaxis of variceal bleed
* Severe cardiopulmonary or renal disease
* Bradycardia (basal heart rate, <50 beats per minute [bpm]) or complete heart block
* A history of severe side effects or contraindications to β- blockers, like bronchial asthma, diabetes mellitus, heart failure, peripheral vascular disease, prostatic hypertrophy, or arterial hypotension (systolic blood pressure <90 mm Hg)
* Refusal to give informed written consent to participate in the trial
* Patients bleeding from gastric varices or Portal Hypertensive Gastropathy (PHG).
* Patients who had a failure of primary hemostasis during acute bleed were also excluded.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Rebleed, death | At least 3 months after last enrollment

SECONDARY OUTCOMES:
Adverse effects of EVL or drug therapy, variceal eradication on EVL, variceal recurrence after eradication on EVL, decrease in variceal grade in the propranolol limb | At least 3 months after last enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — G.B. Pant Hospital, New Delhi, India
Locations (1):
- Department of Gastroenterology, GB Pant Hospital,, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Sarin SK, Gupta N, Jha SK, Agrawal A, Mishra SR, Sharma BC, Kumar A. Equal efficacy of endoscopic variceal ligation and propranolol in preventing variceal bleeding in patients with noncirrhotic portal hypertension. Gastroenterology. 2010 Oct;139(4):1238-45. doi: 10.1053/j.gastro.2010.06.017. Epub 2010 Jun 12. PMID 20547163